CLINICAL TRIAL: NCT02618707
Title: Changes of Lactate Levels During Cardiopulmonary Bypass in Pediatric Undergoing Cardiac Surgery: Possible Early Marker of Morbidity and Mortality
Brief Title: Lactate Levels During Cardiopulmonary Bypass in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Professor (Anesthesiology and Critical Care)- College of Medicine-Assiut University, Assiut University
Other Study IDs: IRB0000871120
Record Dates: First submitted 2015-11-21; First posted 2015-12-01 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Heart Defects, Congenital
Keywords: Lactate; Congenital cardiac defect; CPB; Pediatric
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Lactic Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lactate: Lactate samples will drawn at specific time points within 5 time intervals: before CPB after induction, during cooling on CPB, during rewarming on CPB, immediately after CPB in the operating room, and after admission to the post-operative intensive care unit.
  Interventions: Other: Lactate

INTERVENTIONS:
Other: Lactate — Lactate samples will drawn at specific time points within 5 time intervals: before CPB after induction, during cooling on CPB, during rewarming on CPB, immediately after CPB in the operating room, and after admission to the post-operative intensive care unit.

SUMMARY:
Many variables measured in critically ill patients have been used to estimate severity of disease, prognosticate morbidity and mortality, evaluate costs of treatment, and finally indicate specific treatment and monitor the adequacy of treatment and its timing. It is unlikely that one measurement can replace all of these, but in the remainder of this manuscript the investigators will show that lactate levels may come close. Although in our mind strongly linked to tissue hypoxia, lactate levels follow many more metabolic processes not related to tissue hypoxia and, therefore, subject to many disturbances found in various clinical situations

DETAILED DESCRIPTION:
Forty consecutive pediatric patients who required cardiopulmonary bypass for repair or palliation of complex congenital heart disease will be enrolled in this study. Patients for the study were selected by convenience sampling, without randomization or control of surgical procedure, conduct of anesthesia, or CPB management.

Patients will be monitored intra-operatively using ECG, invasive and non-invasive blood pressure monitoring, pulse oximetry and capnography for determination of End Tidal Co2 ( ETCo2 ) and nasopharyngeal temperature. After induction of anesthesia and placement of an intra-arterial catheter 1 ml of arterial blood will collected into a heparinized 3 ml blood gas syringe and immediately analyzed on the arterial blood gas analyzer (GEM Premier 3000) for blood gas, hematocrit, electrolytes, calcium and glucose. Management strategy of cardio-pulmonary bypass (CPB) was standardized for all the patients. Lactate samples will drawn at specific time points within 5 time intervals: before CPB after induction, during cooling on CPB, during rewarming on CPB, immediately after CPB in the operating room, and after admission to the post-operative intensive care unit.

Differences in lactate levels related to diagnosis will examined. To examine the effect of patient diagnosis and surgical risk on serum lactate level and outcome, the investigators separated patients into surgical risk categories Risk adjustment for congenital heart surgery (RACHS-1). This classification does not include heart transplantation. Patient mortality and the prevalence of postoperative complications for each of the 3 surgical risk categories relative to the change in lactate will examined.

ELIGIBILITY:
Inclusion Criteria:

* age range (1-12 years)
* Usage of cardiopulmonary bypass

Exclusion Criteria:

* chest problems
* Renal problems
* Hepatic problems

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: cardiac surgery for children with congenital heart defects
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Serum lactate during CPB | first 24 hours
  lactate value (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: sayed abd elshafy, MD, Principal Investigator — associate professor
Locations (1):
- Faculty of Medicine, Asyut, Asyut Governorate, Egypt